CLINICAL TRIAL: NCT04858594
Title: Effect of Periodontitis on the Risk of Bloodstream Infection During Intensive Chemotherapy in Patients With Acute Myeloid Leukemia
Brief Title: Study of Periodontitis and Blood Stream Infection in AML Patients Receiving Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: PI left and research was stopped
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2020LS191; HM2020-37 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: BSI; Periodontitis; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Research samples of gingival sulcus fluid, saliva and serum will be collected at baseline. Additionally the blood will be collected weekly through day 28 (or discharge if sooner), and if the patient develops neutropenic fever NF. NF is defined as an oral temperature of ≥100.4°F combined with an absolute neutrophil count (ANC) of ≤0.5x10^9/L^10
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: with Periodontitis: Patients with periodontitis
  Interventions: Other: Planned Chemotherapy
- Arm B: without Periodontitis: Patients without periodontitis
  Interventions: Other: Planned Chemotherapy

INTERVENTIONS:
Other: Planned Chemotherapy — standard oncologic supportive care including antibiotic prophylaxis

SUMMARY:
This is a prospective, observational study to establish the connection between periodontitis and BSI in AML patients planning to receive intensive chemotherapy.

DETAILED DESCRIPTION:
Once eligibility is confirmed, participants will undergo a specialized baseline periodontal examination, gingival sulcus microbiota sampling and saliva sample at baseline before starting chemotherapy.

Patients will be separated into 2 cohorts, with periodontitis (Arm A) and without periodontitis (Arm B). All patients will receive standard oncologic supportive care including antibiotic prophylaxis. Serum samples will be obtained at baseline, at the onset of neutropenic fever, and weekly until day 28 or discharge (whichever sooner).

Study participation will continue during the duration of standard of care chemotherapy for 28 days or until discharge from hospital, whichever later.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of AML, new diagnosis or relapsed/refractory disease
* Planned intensive inpatient chemotherapy, defined as expected hospitalization for 4 weeks or longer
* Sufficient time to perform periodontal examination and treatment by the end of day 1 of chemotherapy without delaying chemotherapy
* Written informed consent prior to performance of any research related activities

Exclusion Criteria:

* Unstable for transfer to the School of Dentistry
* Fever at the time of enrollment
* Documented blood stream infection at the time of enrollment
* Inherited bleeding diathesis
* Periodontitis requiring treatment before starting chemotherapy
* ANC <0.5 x 10^9/L at the time of enrollment
* Unstable for transfer to the School of Dentistry
* Fever at the time of enrollment
* Documented blood stream infection at the time of enrollment
* Inherited bleeding diathesis
* Periodontitis requiring treatment before starting chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study entry is open to adult patients regardless of gender, race or ethnic background. While there will be every effort to seek out and include women and minority patients, the patient population is expected to be similar to that of other relapsed AML studies at the University Of Minnesota
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with Blood stream infections | Day 28 of chemotherapy
  Number of participants experiencing Blood stream infections (BSI) by day 28 of chemotherapy

SECONDARY OUTCOMES:
Number of participants with Neutropenic fever | Day 28 of chemotherapy
  Number of participants experiencing Neutropenic fever (NF) by day 28 of chemotherapy
Number of participants exposed to different antibiotics | Day 28 of chemotherapy
  Number of participants with antibiotic exposure by day 28 of chemotherapy
Length of hospitalization | Day 28 of chemotherapy
  Number of days the patients were hospitalized
Number of participants who died | Day 28 of chemotherapy
  Number of participants who died by day 28 of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States